CLINICAL TRIAL: NCT03233672
Title: Hypofractionated Post-operative IMRT in Prostate Carcinoma: a Phase I/II Study
Brief Title: Hypo-fractionated Postoperative IMRT in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Catholic University of the Sacred Heart (Other); University of Bologna (Other); Howard University (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Iside-PP-2
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Prostate Cancer
Keywords: adjuvant; hypofractionation; IMRT; phase I-II; prostate neoplasms; radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypo-fractionated postoperative IMRT-SIB (Other): All patients underwent combined, intensified and modulated radiotherapy for five days a week with the following doses: 62.5 Gy to the prostate bed and 45 Gy to pelvis nodes in 25 fractions.
  Interventions: Radiation: Hypo-fractionated postoperative IMRT-SIB

INTERVENTIONS:
Radiation: Hypo-fractionated postoperative IMRT-SIB — intensity-modulated radiation treatment with simultaneous integrated boost

SUMMARY:
To report the outcome of hypo-fractionated radiotherapy after radical prostatectomy (RP) for prostate cancer (PCa) using IMRT-SIB. 124 patients with PCa at high risk of relapse after RP or diagnosis of biochemical relapse were included. Patients received 62.5 Gy to the prostate bed (PB) and 45 Gy to pelvis nodes in 25 fractions. Androgen suppressive therapy was prescribed based on NCCN risk categories. Median follow-up was 30 months.

DETAILED DESCRIPTION:
To report the outcome of hypo-fractionated radiation therapy after radical prostatectomy (RP) for prostate cancer (PCa) using intensity-modulated radiation treatment with simultaneous integrated boost (IMRT-SIB).

One hundred and twenty-four patients with PCa at high risk of relapse after RP or diagnosis of biochemical relapse were included in this phase II study (adjuvant: 106 patients, salvage: 18 patients). All patients received 62.5 Gy to the prostate bed (PB) and 45 Gy to pelvis nodes in 25 fractions. Androgen suppressive therapy was prescribed based on NCCN risk categories. Acute and late toxicities were recorded and evaluated according to RTOG (Radiation Therapy Oncology Group) criteria and RTOG-EORTC (European Organization for Research and Treatment of Cancer) scale, respectively.

Median follow-up was 30 months (13-92).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* prior radical prostatectomy with or without lymphadenectomy
* high-risk patients (positive surgical margins, and/or extracapsular extension, and/or seminal vescicle invasion, and/or probability of nodal metastasis > 7% calculated by the Roach formula after pelvic lymph node dissection with ≤ 13 nodes removed, and/or presence of any positive pelvic nodes) or patients with biochemical relapse (initial post-surgery serum PSA equal or above 0.2 ng/mL with a second confirmatory PSA of the same value)
* ECOG performance status 0-1
* adequate bone marrow function (hemoglobin concentration > 8 g/dl, white blood cell count > 3,000/ mm³, platelet count > 75,000/ mm³)
* pre-treatment computed tomography (CT) scan or magnetic resonance imaging (MRI) of the abdomen and pelvis
* bone scan
* informed consent

Exclusion Criteria:

* prior pelvic radiotherapy
* distant metastases
* macroscopic residual tumor
* pelvic or para-aortic nodes at re-evaluation imaging after surgery
* secondary malignancies
* genetic syndromes of hyper-radio-sensitivity
* chronic inflammatory bowel disease
* previously treated with androgen deprivation therapy
* previously treated with chemotherapy for prostate cancer

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-09-18 (Actual); Primary Completion 2010-09-18 (Actual); Study Completion 2014-09-18 (Actual)

PRIMARY OUTCOMES:
incidence of early treatment-emergent adverse events | < 90 days
  adverse events after radiotherapy. Acute side effets were scored according to the Radiation Therapy Oncology Group (RTOG) scale.

SECONDARY OUTCOMES:
Biochemical relapse free survival | 5 years
  Survival free from increase of PSA livel exceeding 0.2 ng/mL for those with post surgical PSA livel of 0.2 ng/mL or lower, and as two consecutive PSA increases for patients with a postsurgical PSA livel of > 0.2 ng/mL
incidence of late treatment-emergent adverse events were assessed with Radiation | 5 years
  Late complications were assessed with delete Radiation Morbidity Scoring Scheme of the RTOG/European Organization for Research and Treatment of Cancer (EORTC)

OTHER OUTCOMES:
First evidence of any pelvic recurrence | 5 years
  First evidence of any pelvic recurrence
Metastasis-free survival | 5 years
  The first evidence of any extrapelvic recurrence of disease

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Study Director — Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine-DIMES, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No